CLINICAL TRIAL: NCT04602845
Title: The Effects of Remimazolam Tosilate Sedation Compared With Midazolam Sedation in Dental Patients: A Double Blind, Prospective , Randomized Controlled Trial
Brief Title: Remimazolam Tosilate Sedation and Midazolam Sedation in Dental Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yang Xudong, Chief of Department of Anesthesiology, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PKUSSIRB-202056102
Record Dates: First submitted 2020-09-10; First posted 2020-10-26 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Sedation Complication; Midazolam; Remimazolam
Keywords: Remimazolam; Midazolam; Sedation
MeSH Terms: interventions — Fentanyl; Flurbiprofen; Midazolam; remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): Drug administration: 50ug fentanyl and 50mg flurbiprofen at the beginning of induction and pre-prepared drugs labeled "inducers", which contained 3 mg/2ml remimazolam.
  Successful sedation is defined as MOAA/S score less than or equal to 4 points during the whole process of the treatment. If MOAA/S score was greater than 4 points, a single dose of Remimazolam (1 mg) is allowed to deepen sedation. if three times of deepen sedation within 15 minutes still can not achieve successful sedation, this progress will define as failure sedation.
  Interventions: Drug: Fentanyl; Drug: Flurbiprofen; Drug: Remimazolam
- Midazolam group (Active Comparator): Drug administration: 50ug fentanyl and 50mg flurbiprofen at the beginning of induction and pre-prepared drugs labeled "inducers", which contained 2.5 mg/2ml midazolam.
  Successful sedation is defined as MOAA/S score less than or equal to 4 points during the whole process of the treatment. If MOAA/S score was greater than 4 points, a single dose of Midazolam (1 mg) is allowed to deepen sedation. if three times of deepen sedation within 15 minutes still can not achieve successful sedation, this progress will define as failure sedation.
  Interventions: Drug: Fentanyl; Drug: Flurbiprofen; Drug: Midazolam

INTERVENTIONS:
Drug: Fentanyl — 50ug Fentanyl intravenously
Drug: Flurbiprofen — 50mg Fentanyl intravenously
Drug: Midazolam — 2.5mg midazolam in 2ml normal saline intravenously
  Arms: Midazolam group
Drug: Remimazolam — 3mg Remimazolam in 2ml normal saline intravenously
  Arms: Remimazolam group

SUMMARY:
Remimazolam Tosilate is a new short-acting benzodiazepines used in sedation. It has the advantages of rapid metabolism, quick recovery without injection pain. This study aims to compared with Midazolam, study whether Remimazolam Tosilate can achieve the same sedation effect with lower side effects on sedation maintenance period, During the recovery period of anesthesia, can Remimazolam Tosilatebe more stable and rapid.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60
2. BMI in 18-30Kg / m2
3. ASA classification I-II level
4. Sign informed consent
5. Patients whose outpatient treatment time less than 1 hour
6. The methods of local anesthesia including: periosteum infiltration method, periodontal ligament injection method, regional nerve block method

Exclusion Criteria:

1. Patients who are allergic to benzodiazepines, opioids, flumazenil or have contraindications
2. Long-term use of benzodiazepines
3. Long-term use of opioids
4. Participate in other clinical trials within 4 weeks
5. Women during pregnancy or breastfeeding
6. Patients who have a history of drug abuse or long-term alcohol abuse
7. Patients who suffer from mental illness or unable to cooperate with the experiment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Success rates of sedation | Day 0
  Success rates for patients who completed outpatient treatment with sufficient depth of sedation, additional sedation medication less than 5 times /15 minutes, and without the need of propofol for further sedation.

SECONDARY OUTCOMES:
Time to reach ideal sedation | Day 0
  Time to reach Modified Observer Assessment of Sedation Score (MOAA/S) ≤ 3 after drug administration
Differences in blood pressure between the two groups | Day 0
  Differences in blood pressure during the operation between the two groups
Differences in heart rate between the two groups | Day 0
  Differences in heart rate during the operation between the two groups
Differences in basic vital signs between the two groups | Day 0
  Differences in blood pressure, heart rate, and BIS at different points during the operation between the two groups
Deepest sedation of MOAA/S | Day 0
  The lowest intraoperative sedation depth of MOAA/S
Deepest sedation of Bispect ral index(BIS) value | Day 0
  The lowest intraoperative sedation depth of BIS value
Recovery of orientation | Day 0
  Time from the end of the treatment to the recovery of orientation
Benzodiazepine dosage | Day 0
  Intraoperative benzodiazepine dosage
Respiratory complication occurrence rate | Day 0
  Respiratory complication including: intraoperative hypoxemia, respiratory depression and other complications in the two groups.
Discharge time | Day 0
  Time to be allowed to discharge after finishing the treatment
The Hopkins Language Learning Test score | Day 0
  The Hopkins Language Learning Test (HVLT-R) score 15 minutes after the end the of the treatment. HVLT-R is a assessment of the patients' language learning condition , this score is from 0 to 30, the more score patients get means the better of patients' Language Learning condition.
Usage rate of flumazenil | Day 0
  If the patients' MOAA/S less than 4 for more than 15 minutes, flumazenil will be used. The usage rate of flumazenil is the number of patients use flumazenil/ the number of all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xudong Yang, MD, Study Chair — Department of anesthesiology of peking university school of stomatology
Locations (2):
- China (2):
  - Peking University Hospital of Stomatology, Beijing, Beijing Municipality
  - Zijian Guo, Haidian, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided